CLINICAL TRIAL: NCT02939963
Title: Comparison of Two Ventilatory Modes During Spontaneous Breathing Trial in Intubated Patients
Brief Title: Ventilation Strategies During Spontaneous Breathing Trial
Acronym: WEANING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0411; 2016-A01172-49 (Other: ANSM Number)
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Insufficiency
Keywords: weaning; mechanical ventilation; work of breathing; automatic tube compensation; pressure support ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATC then pressure support 7 cm H2O PEP 4 cm H2O (Experimental): spontaneous breathing through endotracheal tube with no ventilator support except for ATC
  Interventions: Procedure: ATC then pressure support 7 cm H2O PEP 4 cm H2O
- pressure support 7 cm H2O PEP 4 cm H2O then ATC (Experimental): ventilator is set to pressure support ventilation mode at set pressure 7 cm H2O above PEEP level of 4 cm H2O
  Interventions: Procedure: Pressure support 7 cm H2O PEP 4 cm H2O then ATC

INTERVENTIONS:
Procedure: ATC then pressure support 7 cm H2O PEP 4 cm H2O — spontaneous breathing through endotracheal tube with no ventilator support except for ATC, the patient is connected to the ventilator with pressure support 0 cm H2O and PEP 4 cm H2O during 30 minutes then 30 minutes of basal pressure support then 30 minutes with pressure support 7 cm H2O PEP 4 cm H2O
  Arms: ATC then pressure support 7 cm H2O PEP 4 cm H2O
Procedure: Pressure support 7 cm H2O PEP 4 cm H2O then ATC — 30 minutes with pressure support 7 cm H2O PEP 4 cm H2O then 30 minutes of basal pressure support then 30 minutes with spontaneous breathing through endotracheal tube with no ventilator support except for ATC, the patient is connected to the ventilator with pressure support 0 cm H2O and PEP 4 cm H2O
  Arms: pressure support 7 cm H2O PEP 4 cm H2O then ATC

SUMMARY:
Patients who are intubated and mechanically ventilated for acute respiratory failure in the Intensive Care Unit (ICU) are at some point eligible for weaning. The common way to wean them from mechanical ventilation is to screen criteria for feasibility and, if present, to test feasibility by performing spontaneous breathing trial. This latter can be done either by setting a low pressure support level (expected to compensate the airflow resistance due to endotracheal tube) or by allowing the patient to breathe spontaneously through the tube without any support from the ventilator. Combination of low pressure assistance strategy (7 cm H2O) and positive expiratory pressure (PEP) of 4 cm H2O is the strategy used in our unit. Such a low pressure support level should actually result in a real assistance and, hence this is not the real spontaneous breathing capacity that is tested. Some ICU ventilators offer the option of compensating for the airflow resistance due to endotracheal tube, automatic tube compensation (ATC). Therefore, investigators aimed at comparing in patients ready to wean the usual procedure in our ICU and the ATC mode. In the ATC arm, the patients are breathing spontaneously through the endotracheal tube and are connected to the ventilator set at inspiratory pressure support of 0 cm H2O, PEP 4 cm H2O and ATC on.

Two parallel arms depending on the order of allocation of each mode: pressure support 7 cm H2O + PEP 4 cm H2O then ATC or the opposite. The primary endpoint is the power of the work of breathing. The hypothesis is that the power of the work of breathing is greater in ATC than in the usual procedure, and hence this latter is a real ventilator support.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or more
* intubated and mechanically ventilated for at least 24 consecutive hours
* staying in the medical ICU at the Croix Rousse Hospital, Lyon, France
* pressure support ventilation 10-15 cm H2O, total respiratory rate 25-35 breaths/min, expired tidal volume 6-8 ml/kg predicted body weight
* meeting criteria for spontaneous breathing trial (able to answer simple questions, no ongoing intravenous sedation, norepinephrine ≤ 1 mg/H, dobutamine ≤ 20 mg/h, fraction of inspired oxygen (FIO2 ≤ 50%), PEP ≤ 5 cm H2O, respiratory rate ≤ 35 breaths/min, saturation in oxygen (SpO2) ≥88%)
* under Dräger Evita XL ou V500 ICU ventilator
* agreement to participate from the patient or next of kin

Exclusion Criteria:

* Chronic respiratory failure under long term home oxygen therapy and/or non invasive ventilation before ICU admission
* Tracheotomy
* nasogastric tube contra-indicated
* thoracic tube in place
* no agreement to participate
* under justice protection
* deprived of freedom
* pregnant or breastfeeding
* not affiliated to social insurance
* involved into another study that may interfere with present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
the power of work of breathing | 30 minutes after onset the ventilator strategy
  the work of breathing is measured from the area subtended by the esophageal pressure - lung volume relationship. The power of work of breathing is obtained by multiplying work of breathing by the respiratory frequency and expressed in Joules/min

SECONDARY OUTCOMES:
Respiratory rate | 30 minutes
  the respiratory rate is measured from the airflow tracing
tidal volume | 30 minutes
  integration of airflow over time during expiration
intrinsic PEP | 30 minutes
  deflection in esophageal pressure up to the first zero flow
occlusion pressure at 100 ms | 30 minutes
  measured from the airway pressure at the first 100 ms after airway occlusion
work of breathing per liter | 30 minutes
  work of breathing normalized for 1 liter tidal volume
Distribution of pulmonary ventilation | 30 minutes
  distribution of pulmonary ventilation will be measured by the Pulmovista system

CONTACTS AND LOCATIONS:
Overall Officials: Claude Guerin, Pr, Principal Investigator — Hôpital de la Croix-Rousse
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Guerin C, Terzi N, Mezidi M, Baboi L, Chebib N, Yonis H, Argaud L, Heunks L, Louis B. Low-pressure support vs automatic tube compensation during spontaneous breathing trial for weaning. Ann Intensive Care. 2019 Dec 13;9(1):137. doi: 10.1186/s13613-019-0611-y. PMID 31836913